CLINICAL TRIAL: NCT02231190
Title: A Randomized, Placebo-Controlled, Double-Blind (Sponsor Unblinded) Study to Investigate Protective Effects of GSK1278863 on Eccentric Exercise Induced Muscle Damage in Healthy Male Volunteers
Brief Title: GSK1278863 Effects on Eccentric Exercise-Induced Muscle Damage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200884
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Tendon Injuries
Keywords: muscle soreness; Muscle damage and recovery; muscle function; eccentric exercise
MeSH Terms: conditions — Tendon Injuries; Myalgia | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1278863 (Experimental): Subjects will be given five oral doses of GSK1278863 100 mg (5mg if a low dose is elected for subjects enrolled after interim analysis). The first dose will be administered immediately after completion of eccentric exercise, and then at 4, 8, 24, and 48 hours
  Interventions: Drug: GSK1278863
- Placebo (Placebo Comparator): Subjects will be given five oral doses of Placebo. The first dose will be administered immediately after completion of eccentric exercise, and then at 4, 8, 24, and 48 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1278863 — GSK1278863 will be supplied as oral tablet of strength 100mg, 5mg(5mg if a low dose is elected for subjects enrolled after interim analysis) to be administered with 240 mL of water after end of eccentric exercise
  Arms: GSK1278863
Drug: Placebo — GSK1278863 matching placebo will be supplied as oral tablets for administration with 240 mL of water after end of eccentric exercise
  Arms: Placebo

SUMMARY:
As per non-clinical studies, prolyl hydroxylase inhibitor GSK1278863 can protect muscle from unaccustomed exercise induced muscle damage and enhance functional muscle repair. This study is designed to investigate arm function, pain and other pharmacodynamic (PD) markers after unaccustomed maximal eccentric exercise with concurrent administration of GSK1278863 or placebo. Primary objective of the study is to evaluate the protective effects of GSK1278863 on eccentric exercise induced muscle injury. Subjects will be randomized in a 1:1 ratio (1 subject on GSK1278863 for every 1 subject on placebo). Each subject will be given five oral doses of GSK1278863/placebo in total. The first dose will be administered immediately after completion of eccentric exercise and then 4, 8, 24, and 48 hours later. Subjects will be housed till day 4 in unit and will return for a follow-up visit 7-10 days after discharge. After enrolment of approximately 30 subjects, enrolment will be paused and planned interim analysis will be performed to decide whether to terminate enrolment/study, continue dosing or to reduce the dose to 5 milligrams (mg).

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:
* Males between 18 and 35 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with hemoglobin values outside the normal range should always be excluded from enrolment.
* Body weight >= 70 kilogram (kg) and Body mass index (BMI) within the range 22.0 to 34.0 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <= 1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Corrected QT interval (QTc) < 450 milliseconds (msec) based on single or average QTc value of triplicate values obtained over a brief recording period. The QT correction formula (Fridericia's) used to determine inclusion and discontinuation should be the same throughout the study.
* At least a 1year history of no regular (2-3 times per week) exercise and no heavy exertion within past week, and in the examining physician's opinion the study participant's physical condition/physique is consistent with a history of no regular physical activity for the past year.
* No strenuous exercise involving the arms during the last 10 weeks (e.g., resistance training, rock climbing, rowing, chopping wood, digging, shovelling, sawing).
* The subject is mentally and legally able to comply with the requirements and restrictions of the protocol and has provided signed informed consent prior to participation in any protocol-specific procedures, including Screening procedures.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

Criteria Based Upon Medical History

* History of dizziness or vertigo.
* Uncontrolled hypertension [diastolic blood pressure (BP) >100 millimeter of mercury (mmHg) or systolic BP >170mmHg] at Screening.
* Taking anti-inflammatory, glucocorticoid or other pain medication more than 2 times per week over the previous month.
* Unwilling to abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks for males. One drink is equivalent to 12 grams(g) of alcohol: 12 ounces [360 milliliter (mL)] of beer, 5 ounces (150mL) of wine or 1.5 ounces (45mL) of 80 proof distilled spirits.

* History of drug abuse or dependence within 6 months of the study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* History of peptic ulcer disease or upper gastrointestinal (GI) bleeding within the past 6 months.
* History of thrombosis defined as deep vein thrombosis, stroke, pulmonary embolism or other thrombosis related condition within 3 months prior to Screening.
* History of myocardial infarction or acute coronary syndrome within 3 months prior to Screening.
* History of stroke or transient ischemic attack within 3 months prior to Screening.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of GSK1278863. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue. Examples of conditions that could interfere with hepatic function include Gilbert's syndrome.
* Evidence of active peptic, duodenal or esophageal ulcer disease at Screening OR history of clinically significant GI bleeding within 3 months prior to Screening.
* Subjects with chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease).
* Subjects with a history of symptomatic right heart failure.
* Subjects with Class III or Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* History of proliferative vascular eye disease (e.g., choroidal or retinal disease, such as neovascular age-related macular degeneration, proliferative diabetic retinopathy or macular edema) based upon having had an ophthalmologic exam within 12 months prior to Screening.
* History of risk factors for hypercoagulable state:
* Factor V Leiden (the most common)
* Prothrombin gene mutation
* Deficiencies of natural proteins that prevent clotting (such as antithrombin III, protein C and protein S)
* Recent vascular trauma or surgeryd
* Central venous catheter placement
* Obesity
* Antiphospholipid antibody syndrome
* Myeloproliferative disorders such as polycythemia vera or essential thrombocytosis
* Paroxysmal nocturnal hemoglobinuria
* Nephrotic syndrome
* Active malignancy or diagnosis of malignancy within 5 years prior to Screening (excluding successfully treated basal or squamous cell carcinoma).

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* Screening hemoglobin level > 17.0 grams per deciliter (g/dl).
* Screening Creatine phosphokinase (CPK) > 5xULN.
* Screening serum creatinine >1.10. Other Criteria
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56-day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unwillingness or inability to follow the procedures, or lifestyle and/or dietary restrictions outlined in the informed consent and as directed by site staff.
* Subject is either an immediate family member of a participating Investigator, study coordinator, employee of an Investigator; or is a member of the staff conducting the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2015-06-12 (Actual); Study Completion 2015-06-12 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary contraction (MVC) following eccentric exercise in subjects treated with GSK1278863 or placebo | Up to 72 hours (hrs)
  Muscle strength is a measure of the amount of force produced during a maximal voluntary contraction of the elbow flexors. It will be assessed in the non-dominant arm by a maximal isometric (fixed length) contraction using Cybex ergometer in a seated position after completion of eccentric exercise

SECONDARY OUTCOMES:
Change in MVC following eccentric exercise from pre-eccentric exercise in subjects treated with GSK1278863 or placebo | Up to 72 hrs
  Change in muscle strength from pre-eccentric exercise to completion of eccentric exercise will be assessed
Percent change in MVC following eccentric exercise from pre-eccentric exercise in subjects treated with GSK1278863 or placebo | Up to 72 hrs
  Percent change in muscle strength from pre-eccentric exercise to completion of eccentric exercise will be assessed
Number of subjects with adverse events(AE) | Up to Day 15
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Vital signs assessment as a safety measure | Up to Day 15
  Vital signs includes systolic and diastolic blood pressure, pulse rate and respiratory rate
Electrocardiogram (ECG) assessment as a safety measure | Up to Day 15
  Single 12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, Total cardiac output (QT), and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals
Laboratory parameters assessment as a safety measure | Up to Day 15
  Laboratory parameters include hematology, clinical chemistry, and urinalysis
Change in subject pain assessment using a visual analog scale | Up to 72 hrs
  Arm pain will be assessed for the exercised arm with a visual analog scale on a scale of 0-100 millimeter (mm) during two stimuli; during passive stretching and during MVC contraction, post-exercise and after completion of eccentric exercise
Change in degree of motion and resting arm angle from post-exercise | Up to 72 hrs
  Subjects will be asked to maximally flex their elbow and then maximally extend their elbow, joint angle will be measured using a manual goniometer at maximum flexion and maximum extension. Range of motion will be calculated by subtracting the flexion angle from the extension angle
Composite of PK parameters | Up to Day 2
  PK parameters include maximum observed concentration (Cmax), time of occurrence of Cmax (tmax), and Area under the concentration-time curve from zero (pre-dose) to 24h [AUC(0-24)]

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- See also: Results for study 200884 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200884?search=study&b'study_ids=200884'#rs